CLINICAL TRIAL: NCT01041469
Title: Pilot Study of Auto-immune Abnormalities Associated With Down Syndrome
Acronym: IMMUTRI
Status: Completed | Type: Observational
Sponsor: Institut Jerome Lejeune (Other)
Collaborators: Fondation Jérôme Lejeune (Other)
Responsible Party: Sponsor
Other Study IDs: IJL-IMM-EP10
Record Dates: First submitted 2009-12-30; First posted 2009-12-31 (Estimated); Last update posted 2012-03-22 (Estimated); Status verified 2009-12

CONDITIONS: Down Syndrome With and Without Auto Immune Abnormalities
Keywords: Down syndrome, Humans,Clinical study,Immunity, Autoimmunity,
MeSH Terms: conditions — Down Syndrome; Autoimmune Diseases

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Cross-Sectional
Biospecimen Retention: Samples With DNA — whole blood and white cells
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- with abnormalities: Down syndrome patients presenting with at least one sign of auto immune abnormality
- without abnormality: Down syndrome patients without any sign of recognized auto immune condition

SUMMARY:
The purpose of the study is to identify biological data linked to auto immune abnormalities associated with Down Syndrome.

ELIGIBILITY:
Inclusion Criteria:

* Free and complete trisomy 21
* aged between 8 and 36 years
* biological or clinical signs of auto-immune disorder (group 1)
* no sign of auto-immune disorder (group 2)

Exclusion Criteria:

* any antimitotic or immune depressing treatment during the last 6 months
* Current infectious disease
* Corticosteroid therapy in the last 3 weeks
* pregnancy

Ages: 8 Years to 36 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Study Population: Down syndrome patients followed in a specialized clinic devoted to healthcare of mentally retarded children and adults
Sampling Method: Non-Probability Sample
Enrollment: 72 (Actual)
Dates: Start 2009-11; Study Completion 2010-12 (Actual)

PRIMARY OUTCOMES:
Auto-antibodies dosage | at enrolment
specific lymphocytes populations count | at enrolment

CONTACTS AND LOCATIONS:
Locations (2):
- France (2):
  - Institut Jerome Lejeune, Paris
  - Laboratoire d'Immunologie Biologique (Unité INSERM U580), Paris

REFERENCES:
- [Background] Friedman DL, Kastner T, Pond WS, O'Brien DR. Thyroid dysfunction in individuals with Down syndrome. Arch Intern Med. 1989 Sep;149(9):1990-3. PMID 2528336